CLINICAL TRIAL: NCT00874341
Title: Dose-Response Effect of Fruit and Vegetables on Insulin Resistance in Healthy People Who Are Overweight and at High Risk of Cardiovascular Disease
Brief Title: Effect of Fruit and Vegetables on Insulin Resistance
Acronym: FIRST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Michelle McKinley, Dr Michelle McKinley, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FSA study N02042
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Disease
Keywords: Fruit; Vegetables; Intervention; Insulin resistance; Cardiovascular disease risk; Dose response; High risk of cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention)
- 2 (Active Comparator): 4 portions fruit and vegetables daily for 12 weeks
  Interventions: Other: Fruit and vegetable intervention
- 3 (Active Comparator): 7 portions of fruit and vegetables daily for 12 weeks
  Interventions: Other: Fruit and vegetable intervention

INTERVENTIONS:
Other: Fruit and vegetable intervention — Dose-response effect of fruit and vegetable intake (1-2 vs 4 vs 7 portions per day for 12 weeks)
  Arms: 2; 3

SUMMARY:
Current evidence indicates that fruit and vegetable intake and dietary patterns rich in fruit and vegetables may be associated with reduced insulin resistance and may reduce the risk of the metabolic syndrome. If proven, this relationship may partly explain the inverse association between fruit and vegetable intake and cardiovascular disease risk. There are currently no published dietary interventions that have examined in detail the relationship between fruit and vegetable intake and insulin resistance. There is, however, some preliminary evidence from whole diet interventions that a diet rich in fruit and vegetables may have a beneficial effect on insulin resistance. Evidence to date indicates that an investigation of the direct association between fruit and vegetable intakes and insulin resistance in a carefully controlled intervention study is warranted. This study will investigate the dose-response effect of fruit and vegetable intake on insulin resistance in people who are overweight and at high-risk of CVD using state-of-the-art techniques.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27-35
* CVD risk >20% over 10 years (using the Joint British Society risk assessment tables)
* Low consumers of fruit and vegetables (<2 portions per day)

Exclusion Criteria:

* Diabetes
* Existing CVD
* Food intolerance/sensitivity preventing adherence to a high fruit and vegetable diet
* Subjects taking antioxidant supplements
* Surgery within the last 3 months
* Pregnancy/lactation
* Aspirin
* Subjects following a weight loss diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (two-step euglycaemic-hyperinsulinaemic clamp) | Start and end of 12 week intervention

SECONDARY OUTCOMES:
Self-reported intake of fruit and vegetables (number of portions per day) | Start and end of 12 week intervention
Cardiovascular risk factors | Start and end of 12 week intervention
Biochemical markers of nutritional status | Start and end of 12 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKinley, PhD, Principal Investigator — Queens University Belfast
Locations (2):
- United Kingdom (2):
  - Queen's University Belfast, Belfast, Northern Ireland
  - Royal Victoria Hospital, Belfast

REFERENCES:
- [Result] Wallace IR, McEvoy CT, Hunter SJ, Hamill LL, Ennis CN, Bell PM, Patterson CC, Woodside JV, Young IS, McKinley MC. Dose-response effect of fruit and vegetables on insulin resistance in people at high risk of cardiovascular disease: a randomized controlled trial. Diabetes Care. 2013 Dec;36(12):3888-96. doi: 10.2337/dc13-0718. Epub 2013 Oct 15. PMID 24130354
- [Derived] Wallace IR, McKinley MC, McEvoy CT, Hamill LL, Ennis CN, McGinty A, Bell PM, Patterson CC, Woodside JV, Young IS, Hunter SJ. Serum 25-hydroxyvitamin D and insulin resistance in people at high risk of cardiovascular disease: a euglycaemic hyperinsulinaemic clamp study. Clin Endocrinol (Oxf). 2016 Sep;85(3):386-92. doi: 10.1111/cen.13100. Epub 2016 Jun 13. PMID 27175553
- [Derived] McEvoy CT, Wallace IR, Hamill LL, Neville CE, Hunter SJ, Patterson CC, Woodside JV, Chakravarthy U, Young IS, McKinley MC. Increasing fruit and vegetable intake has no effect on retinal vessel caliber in adults at high risk of developing cardiovascular disease. Nutr Metab Cardiovasc Dis. 2016 Apr;26(4):318-25. doi: 10.1016/j.numecd.2015.10.010. Epub 2015 Nov 14. PMID 27004617
- [Derived] McEvoy CT, Wallace IR, Hamill LL, Hunter SJ, Neville CE, Patterson CC, Woodside JV, Young IS, McKinley MC. Increasing Fruit and Vegetable Intake Has No Dose-Response Effect on Conventional Cardiovascular Risk Factors in Overweight Adults at High Risk of Developing Cardiovascular Disease. J Nutr. 2015 Jul;145(7):1464-71. doi: 10.3945/jn.115.213090. Epub 2015 May 13. PMID 25972532